CLINICAL TRIAL: NCT05393362
Title: Effectiveness of a Cardiac Rehabilitation Program on Biomechanical, Imaging, and Physiological Biomarkers in Elderly Patients With Heart Failure.
Brief Title: Effectiveness of a Cardiac Rehabilitation Program in Elderly Patients With Heart Failure.
Acronym: FUNNEL+
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaga (Other)
Responsible Party: Principal Investigator, Dr. Antonio I Cuesta-Vargas, PhD.Titular Doctor Physiotherapy Department,University of Malaga.Principal Investigator., University of Malaga
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Funnel+ Study
Record Dates: First submitted 2022-05-16; First posted 2022-05-26 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Heart Failure With Preserved Ejection Fraction; Sarcopenia; Frail Elderly Syndrome; Comorbidities and Coexisting Conditions
Keywords: Cardiovascular Rehabilitation; Physical functional performance; Kinematics; Structural; Physiological; Biomarkers; Functional tests; Heart failure
MeSH Terms: conditions — Sarcopenia; Heart Failure | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Randomized crossover clinical trial at the Hospital Regional Universitario of Malaga
Who Masked: Investigator, Outcomes Assessor
Masking Description: The researchers who perform the assessments and analyzes of the data will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cardiac Rehabilitation Program (CR) (Experimental): The CR program will consist of aerobic exercise sessions and strength exercise sessions. The exercises will be individualized after assessing short effort capacities (strength exercise) and long efforts (aerobic exercise). It will be done four days a week, with a minimum of 48 hours between sessions of the same type of exercise. To make progress will be taking a clinical criterion into account, determined by the absence of symptoms derived from HF at the current intensity, and a temporary criterion where provided that the clinical criterion is met, the intensity will be increased every two-three weeks.
  Interventions: Procedure: Cardiac Rehabilitation Program (CR)
- Control Group (CG) (Active Comparator): The control group will receive two education sessions per week for twelve weeks on the complications derived from Heart Failure (HF), functional deterioration, and healthy lifestyle habits.
  Interventions: Behavioral: Control Group (CG)

INTERVENTIONS:
Procedure: Cardiac Rehabilitation Program (CR) — Strength exercises: strengthe exercise will be performed twice a week for 12 weeks, 4-6 series at 60% RM at the beginning of the program, with a progression towards 85% RM in each functional movement at the end of the intervention. The patients will rest for 90 seconds between series and 3 minutes between exercises. Each session has an estimated duration of between 45-60 min.
  Aerobic exercise: aerobic exercise it will be performed twice a week for twelve weeks, between 45-60 min each session of aerobic exercise. It will be developed on a treadmill or cycle ergometer at 50% of HR max at the beginning of the program with a progression towards 80% of HR max at the end, continuously or internally. The Borg scale will prevail over the objective data to adjust the intensity of each patient, Borg = 10/20 or mBorg = 5/10 at the beginning, with progression to Borg = 14/20 or mBorg = 8/10 at the end.
  Other Names: Exercise Group
  Arms: Cardiac Rehabilitation Program (CR)
Behavioral: Control Group (CG) — The control group will receive two education sessions per week for twelve weeks on the complications derived from Heart Failure (HF), functional deterioration, and healthy lifestyle habits.
  Other Names: Health education group
  Arms: Control Group (CG)

SUMMARY:
The main objective of the study is to assess the effectiveness of a cardiac rehabilitation program on functionality, measured by kinematic analysis, cardiorespiratory capacity, and ventricular ejection fraction in elderly patients with heart failure (HF). Other objectives will be; 1) to validate the kinematic analysis as an objective functional assessment that allows performing a functional stratification based on the severity of impairment ("kinematic phenotypes"), as well as to identify those patients who responders or are not responders to the cardiac rehabilitation program; 2) to develop a functional index that includes objective functional parameters, biomechanical biomarkers (heart and musculoskeletal echography) and physiological biomarkers (maximum consumption of oxygen (VO2 max), maximum heart rate (HR max) and blood lactate levels; 3) to analyse the degree of concordance of biomechanical biomarkers with functional tests normally used in clinical practice and with imaging and physiological biomarkers. A randomized, controlled, crossover clinical trial will be carried out at the Hospital Regional Universitario de Málaga. Clinically stable HF patients ≥70 years old will be included. The cardiac rehabilitation program will last 12 weeks and will follow the recommendations of the European Association of Cardiovascular Prevention and Rehabilitation. The patients will perform different functional tests, which will be at baseline, at 3 months and 6 months of follow-up.

DETAILED DESCRIPTION:
Cardiovascular diseases continue to be the main cause of years of life disability-adjusted disability and the leading cause of death, especially in countries with longer life expectancy. Within cardiovascular diseases, Heart Failure (HF) represents a health problem of the first order, with figures of incidence and increasing prevalence associated with the progressive aging of the population and the significant advances in the treatment of chronic diseases associated with HF. HR reaches high morbidity and mortality and is one of the most common reasons for hospital admission common in elderly people, among whom frailty and sarcopenia are commonly associated. All this means that HF has a great impact both at the care level, personal as well as social and economic for public health systems.

HF is a chronic disease characterized by structural cardiac involvement and/or the function that leads to a decrease in cardiac output, which leads to an inability to satisfy the metabolic demands of the organism. Under this circumstance, they end up producing alterations that lead to dyspnea and fatigue, among other manifestations, which functionally limit patients. These patients have a number of characteristics. Distinctive functional characteristics such as reduced aerobic capacity, decreased speed of gait, decreased muscle strength predominantly in the lower limbs, low physical activity, and intolerance to exercise, so they affect the performance of their activities of daily life and their quality of life. These alterations have been associated independently with survival and risk of admission in patients with HF.

In the assessment of physiological biomarkers or cardiovascular functional parameters, maximal oxygen uptake (Peak VO₂) obtained from a cardiopulmonary exercise test (CPET) was considered the reference test to determine cardiovascular functional capacity, exercise tolerance, and prognosis in patients with HF. Various tests have been used useful for the indirect assessment of functionality and prognosis in patients with HR. Among them is the 6-minute walk test (6-MWT), the short battery of physical performance (SPPB), and the Timed Up and Go (TUG) test to evaluate capacity cardiopulmonary and frailty in patients with HF.

Cardiac rehabilitation (CR) is a multidimensional treatment designed to promote changes in lifestyle and physical activity, optimize medical treatment, control risk factors, and address post-developmental social and psychological issues of heart disease. These CR programs have a strong recommendation (Class I) by the guidelines of the European Society of Cardiology (ESC), the American Association of Heart Association (AHA), and the American College of Cardiology (ACC) in the treatment of patients with chronic HF. In addition, it is a cost-effective intervention in HF, since it improves the prognosis by reducing recurrent hospitalizations and health spending, while it has been associated with an increase in survival. They have also shown benefits in the control of cardiovascular risk factors, in anthropometric variables, in blood, physiological (Peak VO₂), and cardiac imaging biomarkers such as ejection fraction ventricular.

However, biomechanical biomarkers, as an objective measure of the functionality of these patients and, therefore, the benefits of the cardiac rehabilitation programs on these biomechanical biomarkers. These biomarkers could make it possible to quantify normal and pathological movements, the degree of deterioration, plan rehabilitation strategies and evaluate the effect of various interventions. Therefore, they could be useful to identify objective parameter functions that could be affected in patients with HF, help to stratify patients with HF based on different levels of functional impairment, in addition, to identify those responders and non-responders to CR programs. To do this, the sensors inertial sensors have been shown to be a precise and reliable method for kinematic evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Subjects older than 70 years.
* Subjects diagnosed with Heart Failure (HF) followed by the Heart Failure Unit.
* Subjects will be able or filling out questionnaires and perform functional tasks;
* Clinical stability.
* Patients receive optimal treatment.

Exclusion Criteria:

* Participants with cardiac pathologies that do not have an HF situation
* Score on the NYHA scale equal to 4.
* Hospitalization in a period of time equal to or less than 3 months.
* Score on the Mini-Mental scale (MMSE) below 24.
* Inability to get up from the chair at least 5 times
* Inability to walk.
* Inability to walk independently without a gait assist device (cane, crutch, or walker).
* Participation in an experimental study where they receive treatment.
* Inability to provide informed consent.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 65 (Actual)
Dates: Start 2023-03-07 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Physiological biomarkers_Cardiopulmonary Exercise Testing (CPET)-(Peak VO2) | Baseline
  Instruments: Cardiopulmonary Exercise Testing at Ciclo-ergometer Measure: the maximum volume of oxygen intake [VO2,(ml/kg/min)]
Physiological biomarkers_Cardiopulmonary Exercise Testing (CPET)-(Peak VO2) | Post intervention_difference (12 weeks after baseline)
  Instruments: Cardiopulmonary Exercise Testing at Ciclo-ergometer Measure: the maximum volume of oxygen intake [VO2,(ml/kg/min)]
Physiological biomarkers_Cardiopulmonary Exercise Testing (CPET)-(Peak VO2) | Follow up (12 weeks after post-intervention)
  Instruments: Cardiopulmonary Exercise Testing at Ciclo-ergometer Measure: the maximum volume of oxygen intake [VO2,(ml/kg/min)]

SECONDARY OUTCOMES:
Physiological biomarkers _Bioelectrical Impedance Analysis (BIA)- (PhA) | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instrument: Nutrilab Bioimpedance device (Akern 2016 with Biatrodes, Akern electrodes) Bioelectrical Phase Angle (PhA) - as derived from equations related to the parameters of BIVA - recently surged as a possible biomarker for patients with HF. Studies provided data about the application of PhA in the clinical management and in the overall risk stratification of HF patients.
Physiological biomarkers _Bioelectrical Impedance Analysis (BIA)- (R) | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instrument: Nutrilab Bioimpedance device (Akern 2016 with Biatrodes, Akern electrodes) Resistance (R, in Ohm)- is related to the amount of body fluids in the sum of intra- (ICW) and extracellular (ECW) water.
Physiological biomarkers _Bioelectrical Impedance Analysis (BIA)- (Xc) | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instrument: Nutrilab Bioimpedance device (Akern 2016 with Biatrodes, Akern electrodes) Reactance (Xc, in Ohm)-is mainly linked to the inner characteristics of the cell membranes.
Physiological biomarkers _Bioelectrical Impedance Analysis (BIA)- (FFM) | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instrument: Nutrilab Bioimpedance device (Akern 2016 with Biatrodes, Akern electrodes) Fat-free mass (FFM, kg)- represents the sum of bone mineral content (BMC) and total lean tissue measurements.
Physiological biomarkers _Bioelectrical Impedance Analysis (BIA)- (FM) | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instrument: Nutrilab Bioimpedance device (Akern 2016 with Biatrodes, Akern electrodes) Fat mass (FM, Kg) - is the total weight of the body minus the weight of any fat measured. This gives an indication of the water, bone, skin, and internal organs as a combined weight.
Physiological biomarkers _Bioelectrical Impedance Analysis (BIA)- (BCM) | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instrument: Nutrilab Bioimpedance device (Akern 2016 with Biatrodes, Akern electrodes) Body cell mass (BCM,Kg) -is the metabolically active cell mass involved in O2 consumption, CO2 production and energy expenditure. BCM measurement has been suggested as a tool for the evaluation of nutritional status. Since BCM is closely related to energy expenditure, it could also represent a good reference value for the calculation of nutrient needs
Physiological biomarkers _Bioelectrical Impedance Analysis (BIA)- (ECW) | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instrument: Nutrilab Bioimpedance device (Akern 2016 with Biatrodes, Akern electrodes) Extracellular water (ECW, L/m) - is the aqueous component that surrounds cells and reflects clinical status in patients with acute or chronic diseases.
Physiological biomarkers _Bioelectrical Impedance Analysis (BIA)- (TBW) | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instrument: Nutrilab Bioimpedance device (Akern 2016 with Biatrodes, Akern electrodes) Total body water (TBW, L/m)- is integral to clinical care. It has significant implications for patient care that include the dosing of medications, assessment and treatment of dehydration, fluid, and energy requirements for parenteral nutrition, and dialysis prescriptions.
Physiological biomarkers _Bioelectrical Impedance Analysis (BIA)- (ECW/TBW) | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instrument: Nutrilab Bioimpedance device (Akern 2016 with Biatrodes, Akern electrodes) Extracellular Water/Total Body Water Analysis (ECW/TBW)-ratio of Extracellular Water(ECW) to Total Body Water(TBW); an important indicator of body water balance. In a healthy state, ECW/TBW ratio should fall within the range 0.360 to 0.390
Physiological biomarkers _Spirometric assessment-(TV) | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instrument: Spirometry device (Spiro USB and MicroRPM, Micro Medical) Tidall Volume (TV)-the amount of air moved in a normal inspiration or exhalation [TV,(mL/Kg)].
Physiological biomarkers _Spirometric assessment-(VC) | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instrument: Spirometry device (Spiro USB and MicroRPM, Micro Medical) Vital Capacity (VC)-The amount of air that is moved in a maximal unforced inspiration or expiration. [VC,(L)].
Physiological biomarkers _Spirometric assessment-(IRV) | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instrument: Spirometry device (Spiro USB and MicroRPM, Micro Medical) Inspiratory reserve volume(IRV)-Difference between the maximum volume that can be breathed in during a normal breath and in a maximal breath [IRV,(L)].
Physiological biomarkers _Spirometric assessment-(ERV) | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instrument: Spirometry device (Spiro USB and MicroRPM, Micro Medical) Inspiratory reserve volume(IRV)-Difference between the maximum volume that can be exhaled in a normal breath and in a maximal breath [ERV,(L)].
Physiological biomarkers _Spirometric assessment-(IC) | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instrument: Spirometry device (Spiro USB and MicroRPM, Micro Medical) Inspiratory Capacity (IC)-The amount of air that can be breathed in after a normal exhalation [IC,(L)].
Physiological biomarkers _Spirometric assessment-(FVC) | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instrument: Spirometry device (Spiro USB and MicroRPM, Micro Medical) Forced Vital Capacity (FVC)-The amount of air moved in a maximal forced inspiration or expiration [FVC,(%)]; [FVC,(L)].
Physiological biomarkers _Spirometric assessment-(FEV1) | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instrument: Spirometry device (Spiro USB and MicroRPM, Micro Medical) Forced Espiratory Volume1, (FEV1)-The amount of air moved in the first second of a forced exhalation; [FEV1,(mL/seg)].
Physiological biomarkers _Spirometric assessment-(PEF) | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instrument: Spirometry device (Spiro USB and MicroRPM, Micro Medical) Peak Espiratory Flow, (PEF)-The maximum amount of air that can be exhaled per second in a forced exhalation.[PEF,(mL/seg)]; [PEF,(%)]
Physiological biomarkers _Spirometric assessment-(MIP) | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instrument: Spirometry device (Spiro USB and MicroRPM, Micro Medical) Maximal inspiratory pressure(MIP)-the pressure generated during maximal inspiratory effort against a closed system.[MIP,(cm H2O)]
Physiological biomarkers _Spirometric assessment-(MEP) | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instrument: Spirometry device (Spiro USB and MicroRPM, Micro Medical) Maximal Espiratory Pressure (MEP)-the pressure generated during maximal espiratory effort against a closed system.[MEP,(cm H2O)]
Physiological biomarkers _Dynamometric assesment-(MDR-Hd-sEMG) | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instrument: High-Density electromyography device (HDEMG) (64-channel EMG amplifier; OT Bioelettronica+) Mean Discharge Rate of Tibialis Anterior Motor Units [MDR-Hd-sEMG,(Hz)].
Physiological biomarkers _Dynamometric assesment-(VC-Hd-sEMG) | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instrument: High-Density electromyography device (HDEMG) (64-channel EMG amplifier; OT Bioelettronica+) Speed of propagation of Tibialis Anterior Motor Units [VC-Hd-sEMG,(m/s)].
Physiological biomarkers _Dynamometric assesment- (F-Iso-FD-din) | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instrument: Dynamometer (J Tech Medical, Powertrack II Commander) Isometric strength in dorsiflexion of the ankle in both limbs during a 5-second maximal test using a digital hand-held dynamometer [F-Iso.FD-din,(N)].
Physiological biomarkers _Dynamometric assesment- (F-Iso-FD-S) | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instrument: S-Type load cell (Biometrics Ltd) Isometric strength in dorsiflexion of the ankle in both limbs tests using S-Type load cell. The signal shall be analysed and processed using the required software. [F-Iso.FD-S].
Physiological biomarkers _Dynamometric assesment-Timed Up and Go (TUG) | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instruments: a long corridor, a chair, a cone and a chronometer Measure: Time (seg) it takes to get up from a chair, walk 3 meters, turn around, return to the chair and sit down again.
Physiological biomarkers _Dynamometric assesment-Six minute walk test (6-MWT) | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instruments: a long corridor and a chronometer Measure: Evaluate the distance (m) a participant can walk for 6 minutes.
Physiological biomarkers _Dynamometric assesment-Short Physical performance Battery (SPPB) | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instruments: a long corridor, a chair, and a chronometer Measure: A set of short tests that time the time it takes to cover a short distance (4 m), repeat 5 times sit-stand up from the chair, and a set of balance tests (feet together, semi-tandem, and tandem). The end result is a score.
Physiological biomarkers_Metabolic biomarkers_Blood lactate | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instruments: Lactate Pro 2 Blood Lactate Analyzer Measure. Blood lactate (mmol/L)
Physiological biomarkers _Cardiopulmonary Exercise Testing (CPET)-(Peak HR) | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instruments: Cardiopulmonary Exercise Testing at Ciclo-ergometer Measure: Peak of Heart Rate [Peak HR,(bpm)].
Physiological biomarkers _Cardiopulmonary Exercise Testing (CPET)-(HRR) | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instruments: Cardiopulmonary Exercise Testing at Ciclo-ergometer Measure: Heart Rate Reserve (HRR)- the difference between the predicted maximal heart rate and the heart rate measured in VO2peak. [HRR,(bpm)].
Physiological biomarkers _Cardiopulmonary Exercise Testing (CPET)-(VO2-VT1) | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instruments: Cardiopulmonary Exercise Testing at Ciclo-ergometer Measure: Ventilatory threshold oxygen consumption (VO2-VT1)- submaximal parameter of cardiorespiratory fitness [VO2-VT1,(mL/min)]
Physiological biomarkers _Cardiopulmonary Exercise Testing (CPET)-(VO2/HR,O2 pulse) | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instruments: Cardiopulmonary Exercise Testing at Ciclo-ergometer Measure: Oxygen pulse [O2 pulse] is the ratio between VO2 (mLO2/min) and heart rate (HR - bpm).
Physiological biomarkers _Cardiopulmonary Exercise Testing (CPET)-(CRE) | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instruments: Cardiopulmonary Exercise Testing at Ciclo-ergometer Measure: Chronotropic Response to Exercise (CRE)-percentage of the chronotropic index [CRE,(%)]
Physiological biomarkers _Cardiopulmonary Exercise Testing (CPET)- (OUES) | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instruments: Cardiopulmonary Exercise Testing at Ciclo-ergometer Measure: Oxygen uptake efficiency slope (OUES)- the ratio of VO2 to the logarithm in base 10 of VE. OUES can be extracted from submaximal tests. [OUES]
Physiological biomarkers _Cardiopulmonary Exercise Testing (CPET)-(RER) | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instruments: Cardiopulmonary Exercise Testing at Ciclo-ergometer Measure: The respiratory exchange ratio [RER] is the ratio of VCO2/VO2
Physiological biomarkers _Cardiopulmonary Exercise Testing (CPET)-(PeakW) | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instruments: Cardiopulmonary Exercise Testing at Ciclo-ergometer Measure: Peak W (Peak work rate)- highest work rate achieved during a maximum of 30 seconds during a stress test [PeakW,(W/min)].
Physiological biomarkers _Cardiopulmonary Exercise Testing (CPET)-(ΔVO2/ΔWR) | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instruments: Cardiopulmonary Exercise Testing at Ciclo-ergometer Measure: [ΔVO2/ΔWR] Relationship. It is defined as the relationship between VO2 (Y-axis in mL.min-1) and workload (X-axis in Watts), measured only during exercise on a cycle ergometer with ramp protocol, whose value is progressively and linearly incremented until maximal effort.
Physiological biomarkers _Cardiopulmonary Exercise Testing (CPET)-(PeakVE) | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instruments: Cardiopulmonary Exercise Testing at Ciclo-ergometer Measure: Peak Pulmonary Ventilation (PeakVE)- highest volume of air moved in and out of the lung [PeakVE,(L/min)]
Physiological biomarkers _Cardiopulmonary Exercise Testing (CPET)-(Vd/Vt) | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instruments: Cardiopulmonary Exercise Testing at Ciclo-ergometer Measure: Physiologic dead space over tidal volume (Vd/Vt) - a routine measurement, expressing the ratio of dead-space ventilation (VD) to tidal ventilation (VT)
Physiological biomarkers _Cardiopulmonary Exercise Testing (CPET)-(VE/MVV) | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instruments: Cardiopulmonary Exercise Testing at Ciclo-ergometer Measure: Breathing reserve [VE/MVV] represents the ratio between maximal ventilation during exercise (VE) and maximum voluntary ventilation (MVV) at rest, both variables in L/min.
Physiological biomarkers _Cardiopulmonary Exercise Testing (CPET)-(PETCO2) | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instruments: Cardiopulmonary Exercise Testing at Ciclo-ergometer Measure: End-tidal CO2 partial pressure [PETCO2, (mmHg)]
Physiological biomarkers _Cardiopulmonary Exercise Testing (CPET)-(PETO2) | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instruments: Cardiopulmonary Exercise Testing at Ciclo-ergometer Measure: End-tidal O2 partial pressure [PETO2, (mmHg)]
Physiological biomarkers _Cardiopulmonary Exercise Testing (CPET)-(VE/VCO2) | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instruments: Cardiopulmonary Exercise Testing at Ciclo-ergometer Measure: Ventilatory equivalents for oxygen [VE/VO2], the ratios between pulmonary ventilation and CO2 production(VE/VCO2)
Physiological biomarkers _Cardiopulmonary Exercise Testing (CPET)-(VE/VO2) | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instruments: Cardiopulmonary Exercise Testing at Ciclo-ergometer Measure: Ventilatory equivalents for oxygen [VE/VO2], the ratios between pulmonary ventilation and O2 consumption (VE/VO2)
Physiological biomarkers_Blood biomarkers_ Complete Blood Cell Count (CBC)_hematocrit | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instruments: The blood test. The extraction of the blood sample must be carried out by a qualified professional (Physician or Nurse). For data analysis, the samples will be sent to the laboratory to recounter de sample.
  Measure: hematocrit (%)
Physiological biomarkers_Blood biomarkers_ Complete Blood Cell Count (CBC)_hemoglobin | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instruments: The blood test. The extraction of the blood sample must be carried out by a qualified professional (Physician or Nurse). For data analysis, the samples will be sent to the laboratory to recounter de sample.
  Measure: hemoglobin 1AC, blood (%)
Physiological biomarkers_Blood biomarkers_ Complete Blood Cell Count (CBC)_Mean Corpuscular Volume (MCV) | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instruments: The blood test. The extraction of the blood sample must be carried out by a qualified professional (Physician or Nurse). For data analysis, the samples will be sent to the laboratory to recounter de sample.
  Measure: mean corpuscular volume [MCV,(fL)]
Physiological biomarkers_Blood biomarkers_ Complete Blood Cell Count (CBC)_Mean Corpuscular Hemoglobin (MCH) | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instruments: The blood test. The extraction of the blood sample must be carried out by a qualified professional (Physician or Nurse). For data analysis, the samples will be sent to the laboratory to recounter de sample.
  Measure: mean corpuscular hemoglobin [MCH,(pg)]
Physiological biomarkers_Blood biomarkers_ Complete Blood Cell Count (CBC)_Mean Corpuscular Hemoglobin Concentration (MCHC) | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instruments: The blood test. The extraction of the blood sample must be carried out by a qualified professional (Physician or Nurse). For data analysis, the samples will be sent to the laboratory to recounter de sample.
  Measure: mean corpuscular hemoglobin [MCHC,(g/dL)]
Physiological biomarkers_Blood biomarkers_ Complete Blood Cell Count (CBC)_Leukocytes | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instruments: The blood test. The extraction of the blood sample must be carried out by a qualified professional (Physician or Nurse). For data analysis, the samples will be sent to the laboratory to recounter de sample.
  Measure: leukocytes (mg/dL)
Physiological biomarkers_Blood biomarkers_ Complete Blood Cell Count (CBC)_Platelet count | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instruments: The blood test. The extraction of the blood sample must be carried out by a qualified professional (Physician or Nurse). For data analysis, the samples will be sent to the laboratory to recounter de sample.
  Measure: platelet count (units/mcL)
Physiological biomarkers_Blood biomarkers_ Complete Blood Cell Count (CBC)_Glomerular Filtration Rate (GFR) | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instruments: The blood test. The extraction of the blood sample must be carried out by a qualified professional (Physician or Nurse). For data analysis, the samples will be sent to the laboratory to recounter de sample.
  Measure: glomerular filtration rate [GFR, (mL/min/1.73m²)]
Physiological biomarkers_Blood biomarkers_ Complete Blood Cell Count (CBC)_Creatinine | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instruments: The blood test. The extraction of the blood sample must be carried out by a qualified professional (Physician or Nurse). For data analysis, the samples will be sent to the laboratory to recounter de sample.
  Measure: creatinine (mg/dL)
Physiological biomarkers_Blood biomarkers_ Complete Blood Cell Count (CBC)_Glucose | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instruments: The blood test. The extraction of the blood sample must be carried out by a qualified professional (Physician or Nurse). For data analysis, the samples will be sent to the laboratory to recounter de sample.
  Measure: glucose (mmol/L)
Physiological biomarkers_Blood biomarkers_ Complete Blood Cell Count (CBC)_Uric Acid | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instruments: The blood test. The extraction of the blood sample must be carried out by a qualified professional (Physician or Nurse). For data analysis, the samples will be sent to the laboratory to recounter de sample.
  Measure: uric acid (mg/dL)
Physiological biomarkers_Blood biomarkers_ Complete Blood Cell Count (CBC)_sodium, potassium, calcium | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instruments: The blood test. The extraction of the blood sample must be carried out by a qualified professional (Physician or Nurse). For data analysis, the samples will be sent to the laboratory to recounter de sample.
  Measure: sodium, potassium, and calcium (mmol/L)
Physiological biomarkers_Blood biomarkers_ Complete Blood Cell Count (CBC)_transaminases -ALT, AST, GGT, FA | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instruments: The blood test. The extraction of the blood sample must be carried out by a qualified professional (Physician or Nurse). For data analysis, the samples will be sent to the laboratory to recounter de sample.
  Measure:transaminases
  * Aminotransferase, alanine [ALT, (U/L)]
  * Aminotransferase, aspartate [AST,(U/L)]
  * Gamma-glutamyl transpeptidase [GGT,(U/L)]
  * Alpha fetoprotein[FA,(mcg/L)]
Physiological biomarkers_Blood biomarkers_ Complete Blood Cell Count (CBC)_glycated hemoglobin | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instruments: The blood test. The extraction of the blood sample must be carried out by a qualified professional (Physician or Nurse). For data analysis, the samples will be sent to the laboratory to recounter de sample.
  Measure: glycated hemoglobin (mmol/mol)
Physiological biomarkers_Blood biomarkers_ Complete Blood Cell Count (CBC)_ferritin | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instruments: The blood test. The extraction of the blood sample must be carried out by a qualified professional (Physician or Nurse). For data analysis, the samples will be sent to the laboratory to recounter de sample.
  Measure: ferritin (ng/mL)
Physiological biomarkers_Blood biomarkers_ Complete Blood Cell Count (CBC)_iron | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instruments: The blood test. The extraction of the blood sample must be carried out by a qualified professional (Physician or Nurse). For data analysis, the samples will be sent to the laboratory to recounter de sample.
  Measure: iron (mcg/dL)
Physiological biomarkers_Blood biomarkers_ Complete Blood Cell Count (CBC)_Index of transferrin saturation | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instruments: The blood test. The extraction of the blood sample must be carried out by a qualified professional (Physician or Nurse). For data analysis, the samples will be sent to the laboratory to recounter de sample.
  Measure: index of transferrin saturation (%)
Physiological biomarkers_Blood biomarkers_ Complete Blood Cell Count (CBC)_transferrin | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instruments: The blood test. The extraction of the blood sample must be carried out by a qualified professional (Physician or Nurse). For data analysis, the samples will be sent to the laboratory to recounter de sample.
  Measure: transferrin (mg/dL)
Physiological biomarkers_Blood biomarkers_ Complete Blood Cell Count (CBC)_ vitamin B12 | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instruments: The blood test. The extraction of the blood sample must be carried out by a qualified professional (Physician or Nurse). For data analysis, the samples will be sent to the laboratory to recounter de sample.
  Measure: vitamin B12 (pg/mL)
Physiological biomarkers_Blood biomarkers_ Complete Blood Cell Count (CBC)_ folic acid | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instruments: The blood test. The extraction of the blood sample must be carried out by a qualified professional (Physician or Nurse). For data analysis, the samples will be sent to the laboratory to recounter de sample.
  Measure: folic acid (ng/mL)
Physiological biomarkers_Blood biomarkers_ Complete Blood Cell Count (CBC)_ HDL | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instruments: The blood test. The extraction of the blood sample must be carried out by a qualified professional (Physician or Nurse). For data analysis, the samples will be sent to the laboratory to recounter de sample.
  Measure: High-density lipoprotein [HDL,(mg/dL)]
Physiological biomarkers_Blood biomarkers_ Complete Blood Cell Count (CBC)_ TSH | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instruments: The blood test. The extraction of the blood sample must be carried out by a qualified professional (Physician or Nurse). For data analysis, the samples will be sent to the laboratory to recounter de sample.
  Measure: TSH (mclU/mL)
Physiological biomarkers_Blood biomarkers_ Complete Blood Cell Count (CBC)_ Total cholesterol (TC) | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instruments: The blood test. The extraction of the blood sample must be carried out by a qualified professional (Physician or Nurse). For data analysis, the samples will be sent to the laboratory to recounter de sample.
  Measure: total cholesterol [TC,(mg/dL)]
Physiological biomarkers_Blood biomarkers_ Complete Blood Cell Count (CBC)_ LDL | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instruments: The blood test. The extraction of the blood sample must be carried out by a qualified professional (Physician or Nurse). For data analysis, the samples will be sent to the laboratory to recounter de sample.
  Measure: Low-density lipoprotein [LDL,(mg/dL)]
Physiological biomarkers_Blood biomarkers_ Complete Blood Cell Count (CBC)_ albumin | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instruments: The blood test. The extraction of the blood sample must be carried out by a qualified professional (Physician or Nurse). For data analysis, the samples will be sent to the laboratory to recounter de sample.
  Measure: albumin (g/dL)
Physiological biomarkers_Blood biomarkers_ Complete Blood Cell Count (CBC)_ triglycerides | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instruments: The blood test. The extraction of the blood sample must be carried out by a qualified professional (Physician or Nurse). For data analysis, the samples will be sent to the laboratory to recounter de sample.
  Measure: triglycerides (mg/dL9
Physiological biomarkers_Blood biomarkers_ Complete Blood Cell Count (CBC)_ NT-proBNP | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instruments: The blood test. The extraction of the blood sample must be carried out by a qualified professional (Physician or Nurse). For data analysis, the samples will be sent to the laboratory to recounter de sample.
  Measure:N-Terminal propeptide of BNP[NT-proBNP,(pg/mL)]
Physiological biomarkers_Blood biomarkers_ Complete Blood Cell Count (CBC)_ vitamin D. | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instruments: The blood test. The extraction of the blood sample must be carried out by a qualified professional (Physician or Nurse). For data analysis, the samples will be sent to the laboratory to recounter de sample.
  Measure: vitamin D (ng/ml)
Biomechanical biomarkers _ RGB-D camera (depth camera)_Trunk linear acceleration | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instruments: RGB-D camera or depth camera. Kinematic analysis by 3D motion capture.
  Measure:
  Trunk linear acceleration (m/s2)
Biomechanical biomarkers_ RGB-D camera (depth camera)_Trunk angular displacement | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instruments: RGB-D camera or depth camera. Kinematic analysis by 3D motion capture.
  Measure:
  Trunk angular displacement (°)
Biomechanical biomarkers _ RGB-D camera (depth camera)_Trunk angular velocity | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instruments: RGB-D camera or depth camera. Kinematic analysis by 3D motion capture.
  Measure:
  Trunk angular velocity (°/s)
Biomechanical biomarkers_ Shimmer3_Step and stride length | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instruments: Inertial sensor (Accelerometer, Gyroscope, and Magnetometer) included in the Shimmer3 instrument.
  Measure:
  Step and stride length
Biomechanical biomarkers_ Shimmer3_Step and stride time | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instruments: Inertial sensor (Accelerometer, Gyroscope, and Magnetometer) included in the Shimmer3 instrument.
  Measure:
  Step and stride time (seg)
Biomechanical biomarkers _ Shimmer3_Step and stride widths stride | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instruments: Inertial sensor (Accelerometer, Gyroscope, and Magnetometer) included in the Shimmer3 instrument.
  Measure:
  Step and stride widths stride
Biomechanical biomarkers _ Shimmer3_Swing phase time gait | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instruments: Inertial sensor (Accelerometer, Gyroscope, and Magnetometer) included in the Shimmer3 instrument.
  Measure:
  Swing phase time gait
Biomechanical biomarkers _ Shimmer3_Gait speed (m/s) | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instruments: Inertial sensor (Accelerometer, Gyroscope, and Magnetometer) included in the Shimmer3 instrument.
  Measure:
  Gait speed (m/s)
Biomechanical biomarkers _ Shimmer3_Stance phase | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instruments: Inertial sensor (Accelerometer, Gyroscope, and Magnetometer) included in the Shimmer3 instrument.
  Measure:
  Stance phase
Biomechanical biomarkers _ Shimmer3_Step speed and stride. | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instruments: Inertial sensor (Accelerometer, Gyroscope, and Magnetometer) included in the Shimmer3 instrument.
  Measure:
  Step speed and stride.
Biomechanical biomarkers _ Shimmer3_Step symmetry | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instruments: Inertial sensor (Accelerometer, Gyroscope, and Magnetometer) included in the Shimmer3 instrument.
  Measure:
  Step symmetry
Imaging biomarkers _Cardiac-Echocardiogram (LVEF) | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instruments: Echocardiogram Measure:Left ventricular Ejection Fraction (%), LVEF
Imaging biomarkers _Cardiac-Echocardiogram (Dilatation and Diameter of the left atrium and left ventricle) | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instruments: Echocardiogram Measure: Dilatation of the left atrium, Dilatation of the left ventricle, Diameter of the left atrium, Diameter of the left ventricle (cm)
Imaging biomarkers _Muscular-Echocardiographic (Muscle Thickness) | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instruments: B-mode ultrasonography device (SonoSite 180 Plus, SonoSite Japan, Tokyo, Japan) Measure: Muscular thickness of the quadriceps rectus muscle ,the diaphragm muscle thickness obtained at the end of inspiration (at total lung capacity; DT-insp) and at resting expiration (at functional residual capacity; DT-exp) through Matlab software (CodigoEco)-[Muscle Thickness]
Imaging biomarkers _Displacement-Echocardiographic (Slide-pL) | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instruments: B-mode ultrasonography device (SonoSite 180 Plus, SonoSite Japan, Tokyo, Japan) Measure: Pleural displacement (Slide-pL, mm) during a complete respiratory cycle through Matlab software (CodigoEco)-[Slide-pL]
Imaging biomarkers_Muscular-Echocardiographic (Fat Thickness) | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instruments: B-mode ultrasonography device (SonoSite 180 Plus, SonoSite Japan, Tokyo, Japan) Measure: Fat thickness of the quadriceps rectus muscle through Matlab software (CodigoEco)-[Fat Thickness]
Imaging biomarkers_Muscular-Echocardiographic (Muscle Echo-Intensity) | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instruments: B-mode ultrasonography device (SonoSite 180 Plus, SonoSite Japan, Tokyo, Japan) Measure: Muscle Echo-intensity of the quadriceps rectus muscle through Matlab software (CodigoEco)- [Muscle His]
Imaging biomarkers_Muscular-Echocardiographic (Fat Echo-Intensity) | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instruments: B-mode ultrasonography device (SonoSite 180 Plus, SonoSite Japan, Tokyo, Japan) Measure: Fat Echo-intensity of the quadriceps rectus muscle through Matlab software (CodigoEco)- [Fat His]
Self-reported_ Borg Rating of Perceived Exertion (RPE)-Borg Scale | Baseline, Post-intervention (12 weeks after baseline) and Follow up (12 weeks after post-intervention)
  Instruments: Borg Rating of Perceived Exertion (RPE)- Borg Scale Measure: The Borg Rating of Perceived Exertion (RPE) is a way of measuring physical activity intensity level. Perceived exertion is how hard you feel like your body is working. It is based on the physical sensations a person experiences during physical activity, including increased heart rate, increased respiration or breathing rate, increased sweating, and muscle fatigue. Although this is a subjective measure, your exertion rating based on a 6 to 20 rating scale, may provide a fairly good estimate of your actual heart rate during physical activity
Self-reported_Sarcopenia Questionnaire (SARC-F) | Baseline, Post-intervention (12 weeks after baseline)
  Instruments: SARC-F questionnaire Measure: It is a simple questionnaire to rapidly diagnose Sarcopenia. It is composed by 5 components: Strength, Assistance to walk, Get up from a chair, Climb stairs and Falls. Scores range from 0 to 10, with 0 to 2 points for each component. A score equal to or greater than 4 could predict sarcopenia and poor results.
Self-reported_abbreviated Comprehensive Geriatric Assessment (aCGA): | Baseline, Post-intervention (12 weeks after baseline)
  Instruments: abbreviated Comprehensive Geriatric Assessment (aCGA): a questionnaire formed by items originating from four different scales.
  Measure: 4 instruments such as:
  * the Geriatric Depression Scale (GDS),
  * the Mini-Mental State Examination (MMSE),
  * Activities of Daily Living (ADL) using the Katz index and instrumental activities of daily living (IADL) using the Lawnton & Brody scale.
  The score varies from 0 to 30 points, giving 1 point to each of the items of the GDS (4 points in total), 12 to the 3 items from the scale of Lawton & Brody, 8 points to the 4 items from the MMSE and 6 points to the 3 items from the Katz index.

OTHER OUTCOMES:
Sociodemographic variables | Baseline
  Instruments: questionnaire, interview.
  Measure:
  * Age
  * Gender
  * Civil Status
  * Educational Level
Anthropometric variables_ Height | Baseline
  Instruments: Weighing machine, measuring tape, calculator Measure: height (cm)
Anthropometric variables_ Weight | Baseline
  Instruments: Weighing machine, measuring tape, calculator Measure: Weight (Kg)
Anthropometric variables_Body Mass Index (BMI). | Baseline
  Instruments: Weighing machine, measuring tape, calculator Measure: body mass index (BMI).
Clinical Variables_Comorbidities | Baseline
  Measure: Comorbidities, specifying number and types Instruments: Comorbidity Index of Charlson
Clinical Variables_Medication | Baseline
  Measure: Medication (specifying number of drugs and types),
Clinical Variables_ Characteristics of the heart failure (HF)_NYHA | Baseline
  Measure: Characteristics of the heart failure (HF) -main cause (ischemic/non-ischemic) Instruments: Grade of the New York Heart Association (NYHA) and symptom score from the Kansas-City questionnaire
Clinical Variables_Hospitalizations in the last 12 months | Baseline
  Measure: Hospitalizations in the last 12 months (number and reason: any cause/HF decompensated),
Clinical Variables_Consultation in the emergency department in the last 12 months | Baseline
  Measure: Consultation in the emergency department in the last 12 months (number and reason: any cause/decompensated HF)
Clinical Variables_Number of falls in the last 12 months | Baseline
  Measure: Number of falls in the last 12 months
Clinical Variables_ Characteristics of the heart failure (HF)_Kansas-City Questionnaire | Baseline
  Measure: Characteristics of the heart failure (HF) -main cause (ischemic/non-ischemic) Instruments: symptom score from the Kansas-City questionnaire
Clinical Variables_Toxic habits | Baseline
  Measure: toxic habits (tobacco, alcohol...).

CONTACTS AND LOCATIONS:
Overall Officials: Cuesta Vargas A Antonio Ignacio, PhD, Principal Investigator — University of Malaga
Locations (1):
- Antonio Cuesta Vargas, Málaga, Spain

REFERENCES:
- [Derived] Cuesta-Vargas AI, Fuentes-Abolafio IJ, Garcia-Conejo C, Diaz-Balboa E, Trinidad-Fernandez M, Gutierrez-Sanchez D, Escriche-Escuder A, Cobos-Palacios L, Lopez-Sampalo A, Perez-Ruiz JM, Roldan-Jimenez C, Perez-Velasco MA, Mora-Robles J, Lopez-Carmona MD, Perez-Cruzado D, Martin-Martin J, Perez-Belmonte LM. Effectiveness of a cardiac rehabilitation program on biomechanical, imaging, and physiological biomarkers in elderly patients with heart failure with preserved ejection fraction (HFpEF): FUNNEL + study protocol. BMC Cardiovasc Disord. 2023 Nov 10;23(1):550. doi: 10.1186/s12872-023-03555-7. PMID 37950216